CLINICAL TRIAL: NCT02457559
Title: An Open-label Study to Assess the Long-term Safety and Efficacy of ONO/GS-4059 in Subjects With Relapsed/Refractory B-cell Malignancies
Brief Title: Study to Assess the Long-term Safety and Efficacy of Tirabrutinib in Adults With Relapsed/Refractory B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-401-1787; 2015-001404-58 (EudraCT Number)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Relapsed/Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence | interventions — tirabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Tirabrutinib 40 mg once daily (CLL) (Experimental): Participants with relapsed/refractory chronic lymphocytic leukemia (CLL) received tirabrutinib 40 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 80 mg once daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 80 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 160 mg once daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 160 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 320 mg once daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 320 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 400 mg once daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 400 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 500 mg once daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 500 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 600 mg once daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 600 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 300 mg twice daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 300 mg twice daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 160 mg once daily (NHL) (Experimental): Participants with relapsed/refractory non-Hodgkin's lymphoma (NHL) received tirabrutinib 160 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 320 mg once daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 320 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 480 mg once daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 480 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 600 mg once daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 600 mg once daily for up to 96 months from first dose in the parent study.
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Tablets or capsules administered orally
  Other Names: ONO/GS-4059

SUMMARY:
The primary objective of this study is to determine the long-term safety and tolerability of tirabrutinib in adults with relapsed/refractory B-cell malignancy who have tolerated and achieved stable disease or improved with tirabrutinib treatment while enrolled in a prior (parent study) tirabrutinib study (NCT01659255). The dosing regimen will be based on the prior dosing regimen from the parent study.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently enrolled in a prior tirabrutinib study
* Did not discontinue treatment with tirabrutinib for any reason other than to enroll in this study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at enrollment in this study
* Any Grade 3 or 4 non-hematologic toxicity that the investigator considers related to previous tirabrutinib use must have resolved, reverted to Grade 1, or reverted to the baseline of the prior study prior to Day 1 of this study
* Negative serum and urine pregnancy test is required for female individuals (unless surgically sterile or greater than 2 years post menopausal)
* Male and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in the protocol
* Lactating females must agree to discontinue nursing before the study drug is administered
* Ability and agreement to attend protocol-specified visits at the study site
* Able to comprehend and willing to sign the informed consent form

Key Exclusion Criteria:

* Known hypersensitivity to tirabrutinib, its metabolites, or formulation excipients

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- France (3):
  - CHRU de Lille, Lille, Nord
  - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - Leicester Royal Infirmary, Leicester
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu H, Truong H, Mitchell SA, Liclican A, Gosink JJ, Li W, Lin J, Feng JY, Jurgensmeier JM, Billin A, Xu R, Patterson S, Pagratis N. Homogeneous BTK Occupancy Assay for Pharmacodynamic Assessment of Tirabrutinib (GS-4059/ONO-4059) Target Engagement. SLAS Discov. 2018 Oct;23(9):919-929. doi: 10.1177/2472555218786165. Epub 2018 Jul 16. PMID 30011241
- [Result] Rule SA, Cartron G, Fegan C, Morschhauser F, Han L, Mitra S, Salles G, Dyer MJS. Long-term follow-up of patients with mantle cell lymphoma (MCL) treated with the selective Bruton's tyrosine kinase inhibitor tirabrutinib (GS/ONO-4059). Leukemia. 2020 May;34(5):1458-1461. doi: 10.1038/s41375-019-0658-7. Epub 2019 Dec 11. No abstract available. PMID 31827243
- [Result] Walter HS, Jayne S, Rule SA, Cartron G, Morschhauser F, Macip S, Karlin L, Jones C, Herbaux C, Quittet P, Shah N, Hutchinson CV, Fegan C, Yang Y, Mitra S, Salles G, Dyer MJS. Long-term follow-up of patients with CLL treated with the selective Bruton's tyrosine kinase inhibitor ONO/GS-4059. Blood. 2017 May 18;129(20):2808-2810. doi: 10.1182/blood-2017-02-765115. Epub 2017 Apr 4. No abstract available. PMID 28377400
- [Result] Walter HS, Rule SA, Dyer MJ, Karlin L, Jones C, Cazin B, Quittet P, Shah N, Hutchinson CV, Honda H, Duffy K, Birkett J, Jamieson V, Courtenay-Luck N, Yoshizawa T, Sharpe J, Ohno T, Abe S, Nishimura A, Cartron G, Morschhauser F, Fegan C, Salles G. A phase 1 clinical trial of the selective BTK inhibitor ONO/GS-4059 in relapsed and refractory mature B-cell malignancies. Blood. 2016 Jan 28;127(4):411-9. doi: 10.1182/blood-2015-08-664086. Epub 2015 Nov 5. PMID 26542378
- [Result] Walter HS, Salles GA, Dyer MJ. New Agents to Treat Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jun 2;374(22):2185-6. doi: 10.1056/NEJMc1602674. No abstract available. PMID 27248633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United Kingdom and France. The first participant was screened on 10 September 2015. The last study visit occurred on 30 December 2020.
Pre-assignment Details: 102 participants were screened. Participants must have been enrolled in parent study ONO-4059POE001 (NCT01659255) to be eligible to receive continued access to tirabrutinib in this rollover study. The dosing regimen was based on the prior dosing regimen from the parent study. As pre-specified in the protocol, the data from both the parent and rollover studies were analyzed together for participants in this rollover study.
Groups:
- Tirabrutinib 80 mg Once Daily (CLL): Participants with relapsed/refractory chronic lymphocytic leukemia (CLL) received tirabrutinib 80 mg once daily for up to 96 months from first dose in parent study.
Period: Overall Study
Arm/Group | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Started | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 2
Completed | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 2 | 3 | 7 | 0 | 1 | 2 | 2 | 0 | 3 | 4 | 2
Not completed — Progressive Disease | 1 | 2 | 3 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1
Not completed — Investigator's Discretion | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all enrolled participants who took at least 1 dose of study drug in the study. The data for this study are summarized by integrating the parent (NCT01659255) study data and rollover study data.
Groups:
- Tirabrutinib 160 mg Once Daily (NHL): Participants with relapsed/refractory NHL received tirabrutinib 160 mg once daily for up to 96 months from first dose in the parent study
- Total: Total of all reporting groups
Arm/Group | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL) | Total
Number analyzed (Participants) | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 2 | 29
Age, Categorical [Count of Participants; unit: Participants] — Age was calculated from the date of first study drug administration of the parent study NCT01659255.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 11
    >=65 years | 0 | 3 | 4 | 0 | 1 | 2 | 2 | 0 | 2 | 3 | 1 | 18
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was from the parent study NCT01659255.
  Participants
    Female | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 6
    Male | 1 | 2 | 6 | 2 | 1 | 2 | 1 | 1 | 3 | 2 | 2 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was from the parent study NCT01659255.
  Participants
    Race: White | 2 | 3 | 5 | 2 | 0 | 2 | 2 | 1 | 2 | 4 | 2 | 25
    Race: Other | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was from the parent study NCT01659255.
  Participants
    Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Ethnicity: Not Hispanic or Latino | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 2 | 29
Region of Enrollment [Number; unit: participants] — All Enrolled Analysis Set included all participants enrolled into this study.
  participants
    United Kingdom | 2 | 2 | 3 | 2 | 0 | 2 | 1 | 1 | 2 | 4 | 1 | 20
    France | 0 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (AEs)
Description: Treatment-emergent AEs were defined as one or both of the following:
  * Any AEs with an onset date on or after the study drug start date of parent study and no later than 30 days after permanent discontinuation of study drug in this rollover study;
  * Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose of tirabrutinib up to 36 months in the parent study and up to 61 months in the rollover study
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug in the study. The data for this study are summarized by integrating the parent (NCT01659255) study data and rollover study data. One participant in 600 mg arm (CLL), received 40 mg dose for a longer period of time in parent study. Hence, this participant was included in 40 mg arm in safety analysis set.
Measure: Number; unit: percentage of participants
Groups:
- Tirabrutinib 40 mg Once Daily (CLL): Participants with relapsed/refractory CLL received tirabrutinib 40 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 300 mg Twice Daily (CLL): Participants with relapsed/refractory CLL received tirabrutinib 300 mg twice daily (BID) for up to 96 months from first dose in the parent study.
Arm/Group | Tirabrutinib 40 mg Once Daily (CLL) | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Number analyzed (Participants) | 1 | 2 | 3 | 7 | 2 | 1 | 1 | 2 | 1 | 3 | 4 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Marked Laboratory Abnormalities
Description: Treatment-emergent marked laboratory abnormalities were defined as values that increase from baseline by at least 3 toxicity grades at any postbaseline time point, up to and including the date of the last dose of study drug plus 30. If the relevant baseline laboratory value is missing, any Grade 3 or 4 values observed within the timeframe specified above will be considered treatment-emergent marked abnormalities. Laboratory assessments included tests for Chemistry, Hematology, Coagulation and Urinalysis.
Time Frame: First dose of tirabrutinib up to 36 months in the parent study and up to 61 months in the rollover study
Population: Participants in the Safety Analysis Set were analyzed. The data for this study are summarized by integrating the parent study (NCT01659255) data and rollover study data. One participant in 600 mg arm (CLL), received 40 mg dose for a longer period of time in parent study. Hence, this participant was included in 40 mg arm in safety analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Tirabrutinib 40 mg Once Daily (CLL) | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Number analyzed (Participants) | 1 | 2 | 3 | 7 | 2 | 1 | 1 | 2 | 1 | 3 | 4 | 2
percentage of participants | 100.0 | 100.0 | 66.7 | 71.4 | 100.0 | 100.0 | 100.0 | 50.0 | 0 | 33.3 | 50.0 | 50.0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined per Modified International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria for CLL and Cheson, 2007 criteria for NHL as percentage of participants who achieve partial response (PR) or complete response (CR) in either parent or roll-over study. CLL:CR: lymphocytes (Ly) <4*10^9/L, no lymphadenopathy,normal spleen and liver size,absence of disease, absolute neutrophil count (ANC) >1.5*10^9/L,platelets ≥100*10^9/L, hemoglobin (Hb) >110 g/L,bone marrow at least normocellular for age; PR: ≥2 of these: ≥50% decrease in Ly, lymphadenopathy,size of liver and spleen, bone marrow infiltrates;and ≥1 of these: ANC >1500/μL, platelets ≥100,000/µL, Hb >11g/dL. NHL:CR: complete resolution of all disease-related radiological abnormalities; PR: ≥50% reduction in sum of products (SPD) of the longest diameters (LD) of all index lesions,no new lesions;no increase in size of liver or spleen;persistence of bone marrow involvement in participant who meets other criteria for CR.
Time Frame: Up to 39 months in parent study and up to 60 months in rollover study
Population: Full Analysis Set consisted of all enrolled participants who took at least 1 dose of study drug in the study. The data for this study are summarized by integrating the parent study (NCT01659255) data and rollover study data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Number analyzed (Participants) | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 2
percentage of participants | 100.0 [15.8 to 100] | 100.0 [29.2 to 100] | 100.0 [59 to 100] | 100.0 [15.8 to 100] | 100.0 [2.5 to 100] | 100.0 [15.8 to 100] | 100.0 [15.8 to 100] | 100.0 [2.5 to 100] | 100.0 [29.2 to 100] | 100.0 [39.8 to 100] | 50.0 [1.3 to 98.7]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined per IWCLL 2008 criteria for CLL and Cheson, 2007 criteria for NHL as the interval from first documentation of CR or PR to the earlier of the first documentation of definitive disease progression as assessed by the investigator, or death from any cause in subjects who achieve a response. CLL:CR: Ly <4*10^9/L, no lymphadenopathy, normal spleen and liver size, absence of disease, ANC >1.5*10^9/L, platelets ≥100*10^9/L, Hb >110 g/L, bone marrow at least normocellular for age; PR: ≥2 of these: ≥50% decrease in Ly, lymphadenopathy, size of liver and spleen, bone marrow infiltrates; and ≥1 of these: ANC >1500/μL, platelets ≥100,000/µL, Hb >11 g/dL. NHL:CR: complete resolution of all disease-related radiological abnormalities; PR: ≥50% reduction in SPD of the LD of all index lesions, no new lesions; no increase in size of liver or spleen; persistence of bone marrow involvement in participant who meets other criteria for CR.
Time Frame: From first documentation of CR or PR to the first documentation of disease progression or death from any cause up to 39 months in parent study and up to 60 months in the rollover study
Population: Participants in the Full Analysis Set with available data were analyzed. Participants who achieved a response are included in the analysis. The data for this study are summarized by integrating the parent study (NCT01659255) data and rollover study data.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Number analyzed (Participants) | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 1
months | NA [61.7 to NA] — Not reached due to insufficient number of participants with events. | 27.0 [26.3 to 42.3] | 57.7 [39.8 to NA] — Not reached due to insufficient number of participants with events. | NA [76.6 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | 33.6 [25.7 to 41.4] | NA [33.6 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | 63.2 [23.9 to 63.2] | 71.4 [53.6 to NA] — Not reached due to insufficient number of participants with events. | 37.0 [37.0 to 37.0]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined per IWCLL 2008 criteria for CLL and Cheson 2007 criteria for NHL as the interval from date of the first dose of tirabrutinib on the parent study to the earlier of the first documentation of definitive disease progression as assessed by the investigator, or death from any cause.
  Progressive disease (PD) in CLL: Lymphadenopathy, or appearance of any new lesion/organomegaly, > 50% increase in the size of the liver and/or spleen, Decrease in platelet count or hemoglobin attributable to CLL per IWCLL, Transformation to a more aggressive histology (eg, Richter syndrome).
  PD in NHL: Cheson, 2007: Appearance of new lesion or increase by >50% of previously involved sites from nadir, Transformation to a more aggressive NHL histology.
Time Frame: From first dose of tirabrutinib in the parent study (NCT01659255) to the first documentation of disease progression or death from any cause up to 99 months
Population: Participants in the Full Analysis Set were analyzed. The data for this study are summarized by integrating the parent study (NCT01659255) data and rollover study data.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Number analyzed (Participants) | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 2
months | NA [63.5 to NA] — Not reached due to insufficient number of participants with events. | 44.0 [28.1 to 44.1] | 59.5 [41.6 to NA] — Not reached due to insufficient number of participants with events. | NA [78.5 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | 35.4 [27.6 to 43.3] | NA [39.1 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | 65.0 [25.8 to NA] — Not reached due to insufficient number of participants with events. | 73.2 [57.3 to NA] — Not reached due to insufficient number of participants with events. | NA [38.9 to NA] — Not reached due to insufficient number of participants with events.

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval from date of the first dose of tirabrutinib on the parent study until death from any cause.
Time Frame: From first dose of tirabrutinib in the parent study (NCT01659255) until death from any cause up to 99 months
Population: Participants in the Full Analysis Set were analyzed. The data for this study are summarized by integrating the parent (NCT01659255) study data and rollover study data.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL)
Number analyzed (Participants) | 2 | 3 | 7 | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 2
months | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [44.8 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [40.8 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [65.0 to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events. | NA [NA to NA] — Not reached due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to 39 months in parent study and up to 61months in the rollover study Adverse Events (AE): First dose of tirabrutinib up to 36 months in the parent study and up to 61 months in the rollover study
Description: All-Cause Mortality: All Enrolled Analysis Set:All participants enrolled in GS-US-401-1787.No participant in 40mg group.
  AE:Safety Analysis Set (SAS):All participants who took at least 1 dose of study drug in this study.For analyses based on SAS, participants were grouped according to actual treatment with longest exposure duration in parent and rollover study. 1 participant in 600mg arm (CLL), received 40mg dose for longer period of time in parent study and was included in 40mg group in SAS.
Groups:
- Tirabrutinib 40 mg QD (CLL): Participants with relapsed/refractory chronic lymphocytic leukemia (CLL) received tirabrutinib 40 mg once daily (QD) for up to 96 months from first dose in the parent study.
- Tirabrutinib 80 mg QD (CLL): Participants with relapsed/refractory CLL received tirabrutinib 80 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 160 mg QD (CLL): Participants with relapsed/refractory CLL received tirabrutinib 160 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 320 mg QD (CLL): Participants with relapsed/refractory CLL received tirabrutinib 320 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 400 mg QD (CLL): Participants with relapsed/refractory CLL received tirabrutinib 400 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 500 mg QD (CLL): Participants with relapsed/refractory CLL received tirabrutinib 500 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 600 mg QD (CLL): Participants with relapsed/refractory CLL received tirabrutinib 600 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 300 mg BID (CLL): Participants with relapsed/refractory CLL received tirabrutinib 300 mg twice daily (BID) for up to 96 months from first dose in the parent study.
- Tirabrutinib 160 mg QD (NHL): Participants with relapsed/refractory non-Hodgkin's lymphoma (NHL) received tirabrutinib 160 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 320 mg QD (NHL): Participants with relapsed/refractory NHL received tirabrutinib 320 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 480 mg QD (NHL): Participants with relapsed/refractory NHL received tirabrutinib 480 mg once daily for up to 96 months from first dose in the parent study.
- Tirabrutinib 600 mg QD (NHL): Participants with relapsed/refractory NHL received tirabrutinib 600 mg once daily for up to 96 months from first dose in the parent study.
Arm/Group | Tirabrutinib 40 mg QD (CLL) | Tirabrutinib 80 mg QD (CLL) | Tirabrutinib 160 mg QD (CLL) | Tirabrutinib 320 mg QD (CLL) | Tirabrutinib 400 mg QD (CLL) | Tirabrutinib 500 mg QD (CLL) | Tirabrutinib 600 mg QD (CLL) | Tirabrutinib 300 mg BID (CLL) | Tirabrutinib 160 mg QD (NHL) | Tirabrutinib 320 mg QD (NHL) | Tirabrutinib 480 mg QD (NHL) | Tirabrutinib 600 mg QD (NHL)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2 | 1/3 | 1/7 | 0/2 | 0/1 | 0/2 | 1/2 | 0/1 | 1/3 | 1/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2 | 3/3 | 5/7 | 1/2 | 0/1 | 1/1 | 1/2 | 0/1 | 2/3 | 4/4 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 3/3 | 7/7 | 2/2 | 1/1 | 1/1 | 2/2 | 1/1 | 3/3 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirabrutinib 40 mg QD (CLL) (N=1) | Tirabrutinib 80 mg QD (CLL) (N=2) | Tirabrutinib 160 mg QD (CLL) (N=3) | Tirabrutinib 320 mg QD (CLL) (N=7) | Tirabrutinib 400 mg QD (CLL) (N=2) | Tirabrutinib 500 mg QD (CLL) (N=1) | Tirabrutinib 600 mg QD (CLL) (N=1) | Tirabrutinib 300 mg BID (CLL) (N=2) | Tirabrutinib 160 mg QD (NHL) (N=1) | Tirabrutinib 320 mg QD (NHL) (N=3) | Tirabrutinib 480 mg QD (NHL) (N=4) | Tirabrutinib 600 mg QD (NHL) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H3n2 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tirabrutinib 40 mg QD (CLL) (N=1) | Tirabrutinib 80 mg QD (CLL) (N=2) | Tirabrutinib 160 mg QD (CLL) (N=3) | Tirabrutinib 320 mg QD (CLL) (N=7) | Tirabrutinib 400 mg QD (CLL) (N=2) | Tirabrutinib 500 mg QD (CLL) (N=1) | Tirabrutinib 600 mg QD (CLL) (N=1) | Tirabrutinib 300 mg BID (CLL) (N=2) | Tirabrutinib 160 mg QD (NHL) (N=1) | Tirabrutinib 320 mg QD (NHL) (N=3) | Tirabrutinib 480 mg QD (NHL) (N=4) | Tirabrutinib 600 mg QD (NHL) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Apical granuloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental pulp disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fat tissue increased (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected bite (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 3 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 3 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinobronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 4 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Tension (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethral caruncle (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethritis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5 | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menopause (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02457559/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02457559/SAP_001.pdf